CLINICAL TRIAL: NCT00059332
Title: Field Administration of Stroke Therapy-Magnesium Trial: A Randomized, Double-Blind, Placebo Controlled Trial of Neuroprotective Magnesium Sulfate Therapy for Acute Stroke Initiated Within 2 Hours of Onset by Paramedics in the Field
Brief Title: Field Administration of Stroke Therapy - Magnesium (FAST-MAG) Trial
Acronym: FAST-MAG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jeffrey L. Saver (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Jeffrey L. Saver, Professor of Neurology, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01NS044364 (NIH); U01NS044364 (NIH)
Record Dates: First submitted 2003-04-23; First posted 2003-04-24 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-06

CONDITIONS: Cerebrovascular Accident
Keywords: stroke; brain attack; magnesium sulfate; neuroprotection; prehospital care; emergency medical services
MeSH Terms: conditions — Stroke | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium Sulfate (Experimental): Magnesium sulfate (Mg) was administered intravenously with a 15 minute bolus load followed by a 24 hour infusion. The bolus-loading dose consisted of 4 grams Mg in 54 ml normal saline. The maintenance infusion contained 16 grams Mg diluted in 240 ml 0.9% normal saline, infused at 10 ml/hr for 24 hours. Paramedics in the field initiated the bolus-loading dose, administered at 216 ml/hr over 15 minutes through a rate controlled IV infusion set. The maintenance infusion was initiated in hospital immediately upon completion of the loading dose.
  Interventions: Drug: Magnesium Sulfate
- Normal saline (Placebo Comparator): Normal saline was administered intravenously with a 15 minute bolus load followed by a 24 hour infusion. Paramedics in the field initiated the bolus-loading dose of 54 ml normal saline, administered at 216 ml/hr over 15 minutes through a rate controlled IV infusion set. The maintenance infusion was initiated in hospital immediately upon completion of the loading dose at 10 ml/hr for 24 hours.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Magnesium Sulfate — Paramedics initiate a loading dose of 4 grams magnesium sulfate IV over 15 minutes, followed after hospital arrival by a maintenance infusion of 16 grams magnesium sulfate IV over 24 hours.
  Other Names: MA 135 magnesium sulfate heptahydrate
  Arms: Magnesium Sulfate
Drug: Normal Saline — Paramedics initiate a loading dose of placebo normal saline IV over 15 minutes, followed after hospital arrival by a maintenance infusion of placebo normal saline IV over 24 hours.
  Other Names: SO155 sodium chloride
  Arms: Normal saline

SUMMARY:
The goal of this study is to evaluate the effectiveness and safety of field-initiated magnesium sulfate in improving the long-term functional outcome of patients with acute stroke.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and the leading cause of adult disability in the United States. Each year, more than 750,000 Americans suffer a symptomatic stroke.

Currently, tissue plasminogen activator (rt-PA) is the only approved treatment for acute ischemic stroke; however, its usefulness is limited because most patients cannot reach medical attention within the necessary 3-hour time window. In addition, rt-PA cannot be given in the field because it is contraindicated for treatment of patients with brain hemorrhage.

The purpose of this multi-center, randomized, double-blind trial is to demonstrate that paramedic initiation of the neuroprotective agent magnesium sulfate in the field is an effective and safe treatment for acute stroke. This study will analyze magnesium sulfate, an experimental therapy for stroke, versus placebo among ambulance-transported patients with acute stroke. This trial will also demonstrate that paramedics can safely, effectively, and rapidly start neuroprotective therapies for stroke.

ELIGIBILITY:
Inclusion Criteria:

* Suspected stroke identified by the Los Angeles Prehospital Stroke Screen
* Age 40-95, inclusive
* Last known well time within 2 hours of treatment initiation
* Deficit present for >/= 15 minutes

Exclusion Criteria:

* Coma
* Rapidly improving neurologic deficit
* Pre-existing neurologic, psychiatric, or advanced systemic disease that would confound the neurological or functional outcome evaluations
* Systolic Blood Pressure (SBP) < 90 or > 220
* Known severe renal dysfunction (on dialysis or known chronic creatinine > 3.0)
* Severe respiratory distress (O2 sat < 90% or respiratory rate < 12 or >/= 24)
* Known second or third degree heart block with no pacemaker in place
* Major head trauma in the last 24 hours
* Recent stroke within prior 30 days
* Patient unable to give informed consent and no available on scene consent or assent provider

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2005-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Saver, M.D., Principal Investigator — UCLA School of Medicine, Study Overall Principal Investigator; Sidney Starkman, M.D., Principal Investigator — UCLA Stroke Center, Co-Principal Investigator; Marc Eckstein, M.D., Principal Investigator — Los Angeles City Emergency Medical Service, Co-Principal Investigator; Samuel Stratton, MD, Principal Investigator — Los Angeles and Orange County Emergency Medical Services Agencies, Co-Principal Investigator; Frank Pratt, MD, Principal Investigator — Los Angeles County Emergency Medical Service, Co-Principal Investigator
Locations (1):
- The Clinical Coordinating Center is: UCLA School of Medicine, 710 Westwood Plaza, Los Angeles, California, United States

REFERENCES:
- [Derived] Kazaryan SA, Shkirkova K, Saver JL, Liebeskind DS, Starkman S, Bulic S, Poblete R, Kim-Tenser M, Guo S, Conwit R, Villablanca P, Hamilton S, Sanossian N. The National Institutes of Health Stroke Scale is comparable to the ICH score in predicting outcomes in spontaneous acute intracerebral hemorrhage. Front Neurol. 2024 Jul 1;15:1401793. doi: 10.3389/fneur.2024.1401793. eCollection 2024. PMID 39011360
- [Derived] Liotta EM, Maas MB, Prabhakaran S, Shkirkova K, Sanossian N, Liebeskind DS, Sharma L, Stratton S, Conwit R, Saver JL; FAST-MAG Investigators and Coordinators. Magnesium and Hematoma Expansion in Intracerebral Hemorrhage: A FAST-MAG Randomized Trial Analysis. Stroke. 2024 Feb;55(2):463-466. doi: 10.1161/STROKEAHA.123.043555. Epub 2023 Dec 21. PMID 38126183
- [Derived] Balucani C, Levine SR, Sanossian N, Starkman S, Liebeskind D, Gornbein JA, Shkirkova K, Stratton S, Eckstein M, Hamilton S, Conwit R, Sharma LK, Saver JL. Neurologic Improvement in Acute Cerebral Ischemia: Frequency, Magnitude, Predictors, and Clinical Outcomes. Neurology. 2023 Mar 7;100(10):e1038-e1047. doi: 10.1212/WNL.0000000000201656. Epub 2022 Dec 7. PMID 36878722
- [Derived] Fan S, Jang M, Kim-Tenser M, Shkirkova K, Liebeskind DS, Starkman S, Villablanca JP, Hamilton S, Naidech A, Saver JL, Sanossian N; FAST-MAG Investigators and Coordinators. Effect of Magnesium on Deterioration and Symptomatic Hemorrhagic Transformation in Cerebral Ischemia: An Ancillary Analysis of the FAST-MAG Trial. Cerebrovasc Dis. 2023;52(5):539-542. doi: 10.1159/000528385. Epub 2023 Jan 4. PMID 36599321
- [Derived] Naidech AM, Shkirkova K, Villablanca JP, Sanossian N, Liebeskind DS, Sharma L, Eckstein M, Stratton S, Conwit R, Hamilton S, Saver JL; FAST-MAG Investigators and Coordinators. Magnesium Sulfate and Hematoma Expansion: An Ancillary Analysis of the FAST-MAG Randomized Trial. Stroke. 2022 May;53(5):1516-1519. doi: 10.1161/STROKEAHA.121.037999. Epub 2022 Apr 5. PMID 35380053
- [Derived] Shkirkova K, Wang TT, Vartanyan L, Liebeskind DS, Eckstein M, Starkman S, Stratton S, Pratt FD, Hamilton S, Kim-Tenser M, Conwit R, Saver JL, Sanossian N. Quality of Acute Stroke Care at Primary Stroke Centers Before and After Certification in Comparison to Never-Certified Hospitals. Front Neurol. 2020 Jan 22;10:1396. doi: 10.3389/fneur.2019.01396. eCollection 2019. PMID 32038463
- [Derived] Shkirkova K, Schuberg S, Balouzian E, Starkman S, Eckstein M, Stratton S, Pratt FD, Hamilton S, Sharma L, Liebeskind DS, Conwit R, Saver JL, Sanossian N; FAST-MAG Investigators and Coordinators. Paramedic Global Impression of Change During Prehospital Evaluation and Transport for Acute Stroke. Stroke. 2020 Mar;51(3):784-791. doi: 10.1161/STROKEAHA.119.026392. Epub 2020 Jan 20. PMID 31955642
- [Derived] Shkirkova K, Saver JL, Starkman S, Wong G, Weng J, Hamilton S, Liebeskind DS, Eckstein M, Stratton S, Pratt F, Conwit R, Sanossian N; FAST-MAG Trial Coordinators and Investigators. Frequency, Predictors, and Outcomes of Prehospital and Early Postarrival Neurological Deterioration in Acute Stroke: Exploratory Analysis of the FAST-MAG Randomized Clinical Trial. JAMA Neurol. 2018 Nov 1;75(11):1364-1374. doi: 10.1001/jamaneurol.2018.1893. PMID 30039165
- [Derived] Chung PW, Kim JT, Sanossian N, Starkmann S, Hamilton S, Gornbein J, Conwit R, Eckstein M, Pratt F, Stratton S, Liebeskind DS, Saver JL; FAST-MAG Investigators and Coordinators. Association Between Hyperacute Stage Blood Pressure Variability and Outcome in Patients With Spontaneous Intracerebral Hemorrhage. Stroke. 2018 Feb;49(2):348-354. doi: 10.1161/STROKEAHA.117.017701. Epub 2018 Jan 4. PMID 29301973
- [Derived] Sanossian N, Rosenberg L, Liebeskind DS, Starkman S, Eckstein M, Stratton S, Pratt FD, Hamilton S, Kim-Tenser M, Sharma LK, Restrepo L, Valdes-Suieras M, Conwit R, Saver JL; FAST-MAG Investigators and Coordinators. A Dedicated Spanish Language Line Increases Enrollment of Hispanics Into Prehospital Clinical Research. Stroke. 2017 May;48(5):1389-1391. doi: 10.1161/STROKEAHA.117.014745. Epub 2017 Apr 7. PMID 28389617
- [Derived] Sanossian N, Apibunyopas KC, Liebeskind DS, Starkman S, Burgos AM, Conwit R, Eckstein M, Pratt F, Stratton S, Hamilton S, Saver JL; FAST-MAG (Field Administration of Stroke Therapy-Magnesium) Investigators and Coordinators. Characteristics and Outcomes of Very Elderly Enrolled in a Prehospital Stroke Research Study. Stroke. 2016 Nov;47(11):2737-2741. doi: 10.1161/STROKEAHA.116.013318. Epub 2016 Sep 27. PMID 27679533
- [Derived] Kim DH, Saver JL, Starkman S, Liebeskind DS, Ali LK, Restrepo L, Kim-Tenser M, Valdes-Sueiras M, Eckstein M, Pratt F, Stratton S, Hamilton S, Conwit R, Sanossian N; Field Administration of Stroke Therapy-Magnesium (FAST-MAG) Trial Nurse-Coordinators and Investigators. Enrollment Yield and Reasons for Screen Failure in a Large Prehospital Stroke Trial. Stroke. 2016 Jan;47(1):232-5. doi: 10.1161/STROKEAHA.115.011687. Epub 2015 Dec 10. PMID 26658446
- [Derived] Sanossian N, Liebeskind DS, Eckstein M, Starkman S, Stratton S, Pratt FD, Koenig W, Hamilton S, Kim-Tenser M, Conwit R, Saver JL; FAST-MAG Investigators and Coordinators. Routing Ambulances to Designated Centers Increases Access to Stroke Center Care and Enrollment in Prehospital Research. Stroke. 2015 Oct;46(10):2886-90. doi: 10.1161/STROKEAHA.115.010264. Epub 2015 Aug 11. PMID 26265130
- [Derived] Saver JL, Starkman S, Eckstein M, Stratton SJ, Pratt FD, Hamilton S, Conwit R, Liebeskind DS, Sung G, Kramer I, Moreau G, Goldweber R, Sanossian N; FAST-MAG Investigators and Coordinators. Prehospital use of magnesium sulfate as neuroprotection in acute stroke. N Engl J Med. 2015 Feb 5;372(6):528-36. doi: 10.1056/NEJMoa1408827. PMID 25651247
- See also: The official FAST-MAG Clinical Trial website — http://www.fastmag.info

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Saline | Magnesium Sulfate
Started | 843 | 857
Completed | 840 | 855
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Magnesium Sulfate | Total
Number analyzed (Participants) | 843 | 857 | 1700
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (13.6) | 69 (13.4) | 69 (13.5)
Age, Customized [Number; unit: participants]
  <60 years of age | 239 | 242 | 481
  60-75 years of age | 284 | 278 | 562
  >75 years of age | 320 | 337 | 657
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 367 | 358 | 725
  Male | 476 | 499 | 975
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 206 | 196 | 402
  Not Hispanic or Latino | 637 | 661 | 1298
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 9
  Asian | 62 | 77 | 139
  Native Hawaiian or Other Pacific Islander | 2 | 6 | 8
  Black or African American | 113 | 106 | 219
  White | 661 | 664 | 1325
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Medical History [Number; unit: participants]
  Hypertension | 648 | 671 | 1319
  Diabetes | 188 | 189 | 377
  Hyperlipidimia | 407 | 398 | 805
  Atrial fibrillation | 175 | 194 | 369
  Myocardial infarction | 82 | 94 | 176
  Tobacco use | 158 | 139 | 297
  Alcohol use | 328 | 326 | 654
Prestroke function - Living at home [Number; unit: participants] | 823 | 834 | 1657
Los Angeles Motor Scale at hospital arrival [Mean (Standard Deviation); unit: units on a scale] — The Los Angeles Motor Scale (LAMS) Facial droop (sub score is 0-1) Absent 0 Present 1 Arm drift (sub score range is 0-2) Absent 0 Drifts down 1 Falls rapidly 2 Grip strength (sub score range is 0-2) Normal 0 Weak grip 1 No grip 2 The sub scales are summed to obtain a total score. Total Score Range is 0-5. Lower values on the scale represent better outcomes and Higher values on the scale represent worse outcomes.
  units on a scale | 3.3 (2.2) | 3.4 (2.3) | 3.4 (2.3)
National Institute of Health Stroke Scale (NIHSS) at hospital arrival [Mean (Standard Deviation); unit: units on a scale] — The National Institute of Health Stroke Scale (NIHSS) is a measure of neurologic deficit. Total Score range 0-42, with higher scores indicating greater severity. The 11 domains assessed are:
  1a-c Level of consciousness 2. Best Gaze 3. Visual 4. Facial Palsy 5a. Motor left arm 5b. Motor right arm 6a. Motor left leg 6b. Motor right leg 7. Limb Ataxia 8. Sensory 9. Best Language 10. Dysarthria 11. Extinction and Inattention
  units on a scale | 11.2 (9.8) | 11.5 (9.9) | 11.3 (9.9)
Intravenous tissue plasminogen activator (t-PA) in patients with cerebral ischemia [Number; unit: participants] | 205 | 242 | 447
Final Diagnosis [Number; unit: participants]
  Cerebral Ischemia | 613 | 632 | 1245
  Intracranial Hemorrhage | 192 | 195 | 387
  Cerebrovascular-mimicking condition | 37 | 30 | 67

OUTCOME MEASURES:

1. Primary Outcome: Modified Rankin Scale
Description: Modified Rankin Scales (mRS) is a measure of global disability. Total Scale range is 0-6, with lower values indicating better outcomes.
  0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Time Frame: 3 months after stroke onset
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Normal Saline | Magnesium Sulfate
Number analyzed (Participants) | 843 | 857
units on a scale | 2 [1 to 4] | 2 [1 to 5]
Statistical Analysis 1: Comparison: Normal Saline vs Magnesium Sulfate; For the primary efficacy analysis, data were analyzed to test the null hypothesis that the distribution of scores over all 7 levels of the modified Rankin Scale at Day 90 was identical in the magnesium sulfate and placebo groups, vs. the one-sided alternative that the distribution of scores is shifted lower in the active magnesium sulfate therapy group. The statistic used to test the primary hypothesis was the Cochran-Mantel-Haenszel test statistic stratified by transport vehicle; Test type: Superiority or Other; p = 0.28, Cochran-Mantel-Haenszel

2. Secondary Outcome: Modified Rankin Score of 0 or 1
Description: Minimal or no disability based on the modified Rankin score
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Normal Saline | Magnesium Sulfate
Number analyzed (Participants) | 843 | 857
participants | 311 | 313
Statistical Analysis 1: Comparison: Normal Saline vs Magnesium Sulfate; Test type: Superiority or Other; p = 0.87, Chi-squared; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.81 to 1.20]

3. Secondary Outcome: Modified Rankin Score ≤2
Description: Functional independence based on modified Rankin score
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Normal Saline | Magnesium Sulfate
Number analyzed (Participants) | 843 | 857
participants | 445 | 449
Statistical Analysis 1: Comparison: Normal Saline vs Magnesium Sulfate; Test type: Superiority or Other; p = 0.87, Chi-squared; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.81 to 1.19]

4. Secondary Outcome: NIH Stroke Scale
Description: The National Institute of Health Stroke Scale (NIHSS) is a measure of neurologic deficit. Total Score range 0-42, with higher scores indicating greater severity. The 11 domains assessed are:
  1a-c Level of consciousness 2. Best Gaze 3. Visual 4. Facial Palsy 5a. Motor left arm 5b. Motor right arm 6a. Motor left leg 6b. Motor right leg 7. Limb Ataxia 8. Sensory 9. Best Language 10. Dysarthria 11. Extinction and Inattention
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Normal Saline | Magnesium Sulfate
Number analyzed (Participants) | 843 | 857
units on a scale | 3 [0 to 42] | 3 [0 to 19]
Statistical Analysis 1: Comparison: Normal Saline vs Magnesium Sulfate; Test type: Superiority or Other; p = 0.2760, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Barthel Index
Description: The Barthel Index is a measure of activities of daily living. Total score is calculated by addition of subscale scores. Total score range is 0-100, with higher scores indicating better outcomes. The ten subitems are:
  FEEDING (Subscale range is 0-10) BATHING (Subscale range is 0-5) GROOMING (Subscale range is 0-5) DRESSING (Subscale range is 0-10) BOWELS (Subscale range is 0-10) BLADDER (Subscale range is 0-10) TOILET USE (Subscale range is 0-10) TRANSFERS (Subscale range is 0-15) MOBILITY (Subscale range is 0-15) STAIRS (Subscale range is 0-10)
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Normal Saline | Magnesium Sulfate
Number analyzed (Participants) | 843 | 857
units on a scale | 95 [20 to 100] | 90 [30 to 100]
Statistical Analysis 1: Comparison: Normal Saline vs Magnesium Sulfate; Test type: Superiority or Other; p = 0.3912, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Stroke Impact Scale
Description: The Stroke Impact Scale (SIS) is a measure of stroke-specific quality of life. The scale assesses 8 domains. Scores for each domain range from 0-100, with higher scores indicating better outcomes.
  1. Physical problems
  2. Memory and thinking
  3. Mood and emotions
  4. Communication, reading and understanding
  5. Daily activities
  6. Mobility at home and in the community
  7. Affected hand use
  8. Hobbies and activities participation
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Normal Saline | Magnesium Sulfate
Number analyzed (Participants) | 843 | 857
units on a scale | 65 [5.4 to 91.7] | 67 [11.7 to 91.7]
Statistical Analysis 1: Comparison: Normal Saline vs Magnesium Sulfate; Test type: Superiority or Other; p = 0.3230, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Serious Adverse Events
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Normal Saline | Magnesium Sulfate
Number analyzed (Participants) | 843 | 857
participants | 422 | 439
Statistical Analysis 1: Comparison: Normal Saline vs Magnesium Sulfate; Test type: Superiority or Other; p = 0.95, Chi-squared; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.87 to 1.27]

8. Secondary Outcome: Symptomatic Intracranial Hemorrhage
Time Frame: 3 month
Measure: Number; unit: participants
Arm/Group | Normal Saline | Magnesium Sulfate
Number analyzed (Participants) | 843 | 857
participants | 28 | 18
Statistical Analysis 1: Comparison: Normal Saline vs Magnesium Sulfate; Test type: Superiority or Other; p = 0.12, Chi-squared; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.34 to 1.14]

9. Secondary Outcome: Mortality
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Normal Saline | Magnesium Sulfate
Number analyzed (Participants) | 843 | 857
participants | 131 | 132
Statistical Analysis 1: Comparison: Normal Saline vs Magnesium Sulfate; Test type: Superiority or Other; p = 0.95, Chi-squared; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.76 to 1.29]

ADVERSE EVENTS:
Time Frame: 3 months after stroke onset
Description: A serious adverse event is one that is fatal or life-threatening, is permanently or substantially disabling, requires or prolongs hospitalization, or is a congenital anomaly, cancer or medication overdose, or any event that the treating clinician judges to be a significant hazard, contraindication, side effect, or precaution.
Arm/Group | Normal Saline | Magnesium Sulfate
Serious Adverse Events (participants affected / at risk) | 422/843 | 439/857
Other Adverse Events (participants affected / at risk) | 331/843 | 329/857
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Saline (N=843) | Magnesium Sulfate (N=857)
Anemia (Blood and lymphatic system disorders) | 8 | 12
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 5 | 2
Atrial fibrillation (Cardiac disorders) | 41 | 43
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 3
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 22 | 28
Cardiac arrest (Cardiac disorders) | 18 | 21
Cardiac discomfort (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 10 | 7
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 5 | 4
Myocardial infarction (Cardiac disorders) | 10 | 13
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 4 | 4
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 2
Syncope (Cardiac disorders) | 2 | 1
Torsade de pointes (Cardiac disorders) | 2 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 3 | 4
Arteriovenous malformation (Congenital, familial and genetic disorders) | 2 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 2 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 44 | 45
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 2
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Parotitis (Gastrointestinal disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 1 | 3
Chest pain (General disorders) | 2 | 3
Fatigue (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pelvic mass (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 22 | 36
Sepsis (Infections and infestations) | 12 | 21
Septic shock (Infections and infestations) | 2 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 17 | 7
Urosepsis (Infections and infestations) | 2 | 2
Wound infection (Infections and infestations) | 1 | 1
Accidental poisoning (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 2 | 4
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Device malfunction (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
Coagulation time prolonged (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Maxillofacial sinus neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Primitive neuroectodermal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Agitation (Nervous system disorders) | 1 | 0
Brain compression (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 3 | 1
Brain oedema (Nervous system disorders) | 22 | 16
Carotid artery stenosis (Nervous system disorders) | 2 | 4
Cerebral haemorrhage (Nervous system disorders) | 25 | 39
Cerebral infarction (Nervous system disorders) | 37 | 32
Cerebral ischaemia (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 11 | 4
Complicated migraine (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 4 | 7
Cytotoxic oedema (Nervous system disorders) | 0 | 3
Depressed level of consciousness (Nervous system disorders) | 2 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 19 | 13
Haemorrhagic transformation stroke (Nervous system disorders) | 6 | 2
Headache (Nervous system disorders) | 2 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 9 | 5
Intracranial pressure increased (Nervous system disorders) | 0 | 2
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 3
Loss of consciousness (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 103 | 105
Paraesthesia (Nervous system disorders) | 1 | 1
Sensory disturbance (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 3 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 3 | 1
Transient ischaemic attack (Nervous system disorders) | 9 | 25
Agitation (Psychiatric disorders) | 1 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 2
Confusional state (Psychiatric disorders) | 1 | 3
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Psychosomatic disease (Psychiatric disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Nephritis interstitial (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 2
Renal failure acute (Renal and urinary disorders) | 6 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 34
Epistaxis (Renal and urinary disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 14
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic valve replacement (Surgical and medical procedures) | 0 | 1
Carotid endarterectomy (Surgical and medical procedures) | 4 | 3
Cranioplasty (Surgical and medical procedures) | 1 | 0
Craniotomy (Surgical and medical procedures) | 5 | 2
Endotracheal intubation (Surgical and medical procedures) | 0 | 1
Haematoma evacuation (Surgical and medical procedures) | 2 | 2
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Lung lobectomy (Surgical and medical procedures) | 1 | 0
Medical device implantation (Surgical and medical procedures) | 0 | 1
Mitral valve replacement (Surgical and medical procedures) | 0 | 1
Transfusion (Surgical and medical procedures) | 1 | 0
Ventricular drainage (Surgical and medical procedures) | 2 | 2
Aortic aneurysm (Vascular disorders) | 1 | 0
Carotid artery dissection (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 31 | 36
Gangrene (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 30 | 59
Malignant hypertension (Vascular disorders) | 1 | 0
Neurogenic shock (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 3
Peripheral vascular disorder (Vascular disorders) | 2 | 1
Syncope (Vascular disorders) | 0 | 2
Vasospasm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=843) | Magnesium Sulfate (N=857)
Headache (General disorders) | 167 (173) | 178 (184)
Hypokalaemia (Blood and lymphatic system disorders) | 214 (233) | 205 (217)
Urinary tract infection (Renal and urinary disorders) | 133 (142) | 138 (152)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No